CLINICAL TRIAL: NCT01884077
Title: Total vs. Reverse Shoulder Replacement: a Prospective Randomized Trial
Brief Title: Total vs. Reverse Shoulder Replacement: Pain Relief Two Years After Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment and poor follow up
Sponsor: Washington University School of Medicine (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201209102
Record Dates: First submitted 2013-06-12; First posted 2013-06-21 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Arthritis
Keywords: patient outcomes two years after shoulder replacement; seventy years of age and older
MeSH Terms: conditions — Arthritis | interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reverse Shoulder Arthroplasty (Active Comparator): Shoulder Joint Replacement Reverse Arthroplasty Implant to surgically replace arthritic shoulder
  Interventions: Device: Total Shoulder Arthroplasty
- Total Shoulder Arthroplasty (Active Comparator): Shoulder Joint Replacement Total Arthroplasty Implant used to surgically replace osteoarthritic shoulder joint
  Interventions: Device: Reverse Shoulder Arthroplasty

INTERVENTIONS:
Device: Reverse Shoulder Arthroplasty — REVERSE In a Reverse Total shoulder the ball is located on the shoulder blade (glenoid) and the socket is located on the arm bone (humerus), exactly the opposite of the situation in a conventional total shoulder. The ball (glenosphere) is screwed to the bone of the shoulder blade. The cup (humeral sock¬et) is fixed to a stem that is cemented down the inside of the arm bone (humerus).
  Arms: Total Shoulder Arthroplasty
Device: Total Shoulder Arthroplasty — TOTAL In a conventional Total shoulder, the arthritic surface of the ball is replaced with a metal ball with a stem that is press fit in the inside of the arm bone (humerus) and the socket is resurfaced with a component.
  Arms: Reverse Shoulder Arthroplasty

SUMMARY:
Specific Aim: To compare early postoperative pain relief in patients over the age of 70 who undergo either Total Shoulder Arthroplasty or Reverse Shoulder Arthroplasty in treatment of glenohumeral osteoarthritis.

Hypothesis: Early postoperative pain relief will be greater in those undergoing Reverse Shoulder Arthroplasty.

DETAILED DESCRIPTION:
The shoulder is the most mobile joint in the human body with a complex arrangement of structures working together to provide the movement necessary for daily life. Great mobility comes at the expense of stability. Several bones and a network of soft tissue (ligaments, tendons, and muscles) work together to produce shoulder movement. They also interact to keep the joint in place while it moves through extreme ranges of motion.

BONES The glenohumeral joint (shoulder joint) is a multiaxial, synovial ball and socket joint and involves articulation between the shoulder blade and the head of the humerus (upper arm bone). This makes it the most mobile joint of the human body.

SOFT TISSUE The rotator cuff is a group of muscles and their tendons that act to stabilize the shoulder. The four muscles of the rotator cuff are over half of the seven scapulohumeral muscles. These tendons can become torn following a trauma to the shoulder or it can occur through the "wear and tear" on tendons, most commonly the supraspinatus tendon found under the acromion. To be considered an equal candidate for both implants the rotator cuff must be grossly intact.

ARTHRITIS Glenohumeral (shoulder) arthritis is a common source of pain and disability that affects up to 20% of the older population. Damage to the cartilage surfaces of the glenohumeral joint (the shoulder's "ball-and-socket" structure) is the primary cause of shoulder arthritis.

SHOULDER REPLACEMENTS There are two types of total shoulder replacement systems: the conventional Total shoulder and the Reverse shoulder. The reverse was originally developed for use in patients with advanced high loss of shoulder function in conjunction with a damaged rotator cuff.

TOTAL In a conventional Total shoulder, the arthritic surface of the ball is replaced with a metal ball with a stem that is press fit in the inside of the arm bone (humerus) and the socket is resurfaced with a component.

REVERSE In a Reverse Total shoulder the ball is located on the shoulder blade (glenoid) and the socket is located on the arm bone (humerus), exactly the opposite of the situation in a conventional total shoulder. The ball (glenosphere) is screwed to the bone of the shoulder blade. The cup (humeral sock¬et) is fixed to a stem that is cemented down the inside of the arm bone (humerus). This configuration provides sta¬bility because the muscles around the shoulder compress the ball and socket together.

STUDY PROCEDURES Randomization to either a total or reverse shoulder replacement Review of medical records and imaging related to patient's shoulder arthritis and surgery Range of motion and strength testing at enrollment and two years post op Completion of American Shoulder & Elbow Survey and WOOD at enrollment and two years post op

There are clear clinical indications for the use of the total and reverse shoulder replacements in patients younger than 70 years old and they are based on cuff integrity and shoulder function. However, the decision to use the total shoulder implant or the reverse total shoulder implant in patients over 70 yrs old with end-stage glenohumeral (shoulder) arthritis and an intact rotator cuff is based on surgeon's preference. There are no studies comparing pain relief for these two implants in this patient population. So this study will randomize 34 patients to either total or reverse shoulder replacements. These individuals must meet the clinical criteria to be a candidate for either implant.

The Reverse Shoulder Arthroplasty has revolutionized the management of complex shoulder pain and dysfunction due to rotator cuff tear arthropathy since its FDA approval in 2003. The indications for the use of the Reverse Shoulder Arthroplasty continue to expand and early results are encouraging for patients with arthritis in the setting of a massively torn rotator cuff. However, the role of the Reverse Shoulder Arthroplasty to manage pain secondary to osteoarthritis of the shoulder in the setting of an intact rotator cuff with underlying age-related rotator cuff degeneration is not clear and remains a challenging clinical question. This question continues to gain significance as the number of patients with shoulder arthritis is rapidly growing as is the number of arthroplasty procedures performed annually.

Glenohumeral (shoulder) arthritis occurs when the normally smooth joint surfaces of glenoid and the humeral head are damaged by congenital, metabolic, traumatic, degenerative, vascular, septic or aseptic inflammatory factors. The prevalence of Glenohumeral arthritis increases with age.1-3 Several studies have evaluated for the prevalence of Glenohumeral arthritis and found that it can be found in up to 16% of the elderly population.4-7 Arthritis of the shoulder has been reported to be a source of severe disability and limitation of the quality of life of those who experience it.8, 9

End stage shoulder arthritis is reliably treated with shoulder arthroplasty. The shoulder is the third most common joint in the body that is replaced. The incidence of shoulder arthroplasty procedures (including hemiarthroplasty, total shoulder arthroplasty and reverse shoulder arthroplasty) is increasing steadily in the United States.10 In 1998 approximately 19,000 shoulder arthroplasty procedures were performed. In 2008 approximately 47,000 shoulder arthroplasty procedures were performed. The incidence of total shoulder arthroplasty has steadily outpaced that of hemiarthroplasty as the preferred choice for management of osteoarthritis. The Reverse shoulder arthroplasty was approved by the FDA in 2003 and since then has steadily gained in popularity. As the elderly population continues to grow and arthroplasty techniques evolve, the number of shoulder arthroplasty performed annually is expected to continue to increase.

Total shoulder arthroplasty relies on an intact and functioning rotator cuff in order to keep the prosthetic head centered on the prosthetic glenoid. Rotator cuff deficiency has been associated with early glenoid component loosening after total shoulder arthroplasty resulting in shoulder pain, dysfunction and revision arthroplasty surgery.8, 11 Rotator cuff degeneration is also associated with advancing age.12

The scenario of age-associated rotator cuff degeneration in conjunction with chronic osteoarthritis is a common clinical presentation. The shoulder with chronic osteoarthritis in the setting of a degenerative or atrophic rotator cuff presents a challenging clinical question. From a management standpoint the question arises of whether the patient would be best served with a total shoulder arthroplasty or a reverse shoulder arthroplasty. A total shoulder arthroplasty is the gold standard arthroplasty option but requires an intact and functional rotator cuff to function properly and an elderly patient is more likely to have rotator cuff degeneration and dysfunction. Rotator cuff dysfunction may be revealed early after undergoing a total shoulder arthroplasty and range of motion improves. Secondary rotator cuff dysfunction after total shoulder arthroplasty is becoming an increasingly recognized entity and clinical challenge.13 Conversely, a reverse shoulder arthroplasty does not require a functional rotator cuff and has been noted to have promising results but is an arthroplasty option with less predictable outcomes and less clinical follow-up.

Many studies have been published that discuss patient outcomes after shoulder arthroplasty.8, 14-17 These studies are limited by small patient populations, limited follow-up, and heterogeneity of patient populations and surgical indications. No study has compared Total Shoulder Arthroplasty with Reverse Shoulder Arthroplasty in the treatment of osteoarthritis in the population older than 70 years of age. The Shoulder and Elbow service at Washington University is uniquely qualified to conduct a study of this type given the exceptionally large surgical volume of shoulder arthroplasty (over 350 shoulder arthroplasty cases performed annually), access to Ultrasonography for imaging of all study participants and a robust and well-organized research infrastructure that can execute established research protocols.

ELIGIBILITY:
Inclusion Criteria:

* age 70 or older,
* have radiographic signs of osteoarthritis (narrowing of the glenohumeral joint space, marginal osteophytes around the humeral head, progressive changes with sclerosis and subcortical cystic formation and flattening of the humeral head),
* intact rotator cuff but with atrophy or fatty degeneration (defined as Grade II atrophy noted on preoperative shoulder ultrasound),
* objective weakness as measured with Isobex testing,
* limited forward elevation (less than 90 degrees)

Exclusion Criteria:

* patients who present with pain secondary to inflammatory arthropathy,
* obvious full-thickness rotator cuff tear,
* cuff tear arthropathy,
* revision arthroplasty,
* fracture or trauma,
* patients who had previous rotator cuff repair or prior open surgery prior to shoulder arthroplasty.
* pregnancy

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01-28 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Chamberlain, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reverse Shoulder Arthroplasty | Total Shoulder Arthroplasty
Started | 8 | 11
Completed | 0 | 1
Not Completed | 8 | 10
Not completed — screen fail | 0 | 2
Not completed — canceled surgery | 2 | 0
Not completed — Lost to Follow-up | 0 | 4
Not completed — study closed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reverse Shoulder Arthroplasty | Total Shoulder Arthroplasty | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 8 | 11 | 19
Age, Continuous [Median (Full Range); unit: years] | 72 [69 to 75] | 77 [72 to 82] | 75.5 [69 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: ASES Score
Description: American Shoulder & Elbow Survey (ASES): Assessment of patient-rated shoulder pain and function/disability. Questions involve activities of daily living that reflect the use of the shoulder & elbow in different planes of motion. Pain and weakness with various activities are also addressed. ASES score will be calculated, compared and reported for both groups pre-operatively and 2 years post operatively: (17 patients) total arthroplasty and (17 patients) reverse arthroplasty.
Time Frame: 2 years after shoulder replacement
Population: This study has been discontinued and data was not sufficiently collected for any participant.
Arm/Group | Reverse Shoulder Arthroplasty | Total Shoulder Arthroplasty
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: WOOS Score
Description: a disease-specific quality-of-life instrument (Western Ontario Osteoarthritis of the Shoulder [WOOS]. WOOS Score will be generated for both groups pre-operatively and 2 years post operatively: Reverse arthroplasty(17 patients) and Total arthroplasty (17 patients)
  Study has been discontinued
Time Frame: 2 years after shoulder replacement
Population: This study has been discontinued. This study has been discontinued and data was not sufficiently collected for any participant.
Arm/Group | Reverse Shoulder Arthroplasty | Total Shoulder Arthroplasty
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Shoulder Strength and Motion Based on Physican Examination
Description: Research team member measures both shoulder range of motion (using a goniometer) and strength based on the standardized American Shoulder and Elbow Surgeons Society (ASES)examination. Physical Examination includes the following: forward elevation, external rotation, internal rotation, external rotation at side, Internal rotation extension with lift off exam, Horn Blower's, external rotation strength, thumb down abduction strength, abdominal compression test, Biceps rupture, Speeds Test, and Yergason's Test. External and Thumb Down abduction are measured with Iso-Force machine. Preoperative and 2 year post-operative range of motion and strength measurement score averages will be compared and reported for both groups (total 34 patients).
Time Frame: 2 years post shoulder replacement
Population: as for outcome 2
Arm/Group | Reverse Shoulder Arthroplasty | Total Shoulder Arthroplasty
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3.5 years
Description: No adverse events
Arm/Group | Reverse Shoulder Arthroplasty | Total Shoulder Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

LIMITATIONS AND CAVEATS:
This study was terminated due to slow enrollment and poor follow up. There is insufficient data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No